CLINICAL TRIAL: NCT07052591
Title: The Effect of Zumba Exercise on Body Composition, Strength, and Balance Skills in Folk Dancers: A Randomized Controlled Trial
Brief Title: The Effect of Zumba Exercise on Body Composition, Strength and Balance Skills in Folk Dancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Ebru CEVİZ (Other)
Responsible Party: Sponsor-Investigator, Dr. Ebru CEVİZ, Assistant Professor, Bingol University
Organization: Bingol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: E-33117789-300-159280
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Body Composition; Muscle Strength; Balance; Healthy Volunteers - Male and Female
Keywords: Zumba; body composition; strength; balance; performance
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned into two parallel groups: an experimental group that performed Zumba exercise sessions twice a week for 8 weeks, and a control group that did not receive any exercise intervention. Both groups underwent pre-test and post-test assessments to evaluate changes in body composition, muscle strength, and balance.
Who Masked: Outcomes Assessor
Masking Description: No masking was applied in this study; both participants and researchers were aware of the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zumba Exercise Group (Experimental): Participants in this arm performed 60-minute Zumba exercise sessions twice per week for 8 weeks. The intervention consisted of aerobic dance routines designed to improve body composition, muscular strength, and balance. All sessions were conducted under the supervision of trained instructors.
  Interventions: Behavioral: Zumba Exercise
- Control Group (Other): Participants in this arm did not receive any structured exercise intervention. They continued their usual daily activities throughout the 8-week study period. No physical training or behavioral program was applied.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Zumba Exercise — Participants in the Zumba Exercise group engaged in supervised aerobic dance sessions lasting 60 minutes, twice per week, over an 8-week period. The exercise intensity was set to match aerobic-level activity suitable for improving body composition, muscle strength, and balance. Sessions included warm-up, main Zumba dance routines, and cool-down phases, all conducted by certified instructors.
  Arms: Zumba Exercise Group
Other: Control Group — Participants in this arm did not receive any structured exercise intervention. They continued their usual daily activities throughout the 8-week study period. No physical training or behavioral program was applied.
  Arms: Control Group

SUMMARY:
This study investigates the effects of an 8-week Zumba exercise program on body composition, muscle strength, and balance skills in male and female folk dancers aged 19-25 years. Participants are randomly assigned to either a Zumba exercise group, performing sessions twice a week, or a control group without exercise. The study aims to determine whether Zumba can improve physical fitness and postural control in folk dancers, especially examining any differences between genders.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the impact of an 8-week aerobic-level Zumba exercise program on body composition, muscle strength, and balance in folk dancers aged 19 to 25 years. Forty-eight participants were randomly assigned into experimental and control groups, with equal numbers of males and females in each. The experimental group participated in 60-minute Zumba sessions twice weekly at predetermined intensity levels, while the control group maintained their usual activities without structured exercise. Outcome measures included body fat percentage, muscle mass ratio, static hand, leg, and back strength, and both static and dynamic balance assessments. The study investigates gender-specific responses to the exercise intervention and seeks to provide evidence on the efficacy of Zumba as a fitness modality for folk dancers.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 19 and 25 years.
* Male and female folk dancers.
* Healthy individuals without any chronic illness or injury that would prevent participation in physical exercise.
* Willingness to participate in the study and provide informed consent.

Exclusion Criteria:

* Presence of any musculoskeletal or neurological disorder affecting balance or strength.
* Participation in other regular physical training programs during the study period.
* Any medical condition contraindicating aerobic exercise.

Ages: 19 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Body Composition | 8 weeks
  Changes in body fat percentage and muscle mass ratio measured before and after the 8-week intervention using bioelectrical impedance analysis.
Muscle Strength | 8 weeks
  Assessment of static hand, leg, and back strength before and after the intervention using standardized strength tests.
Balance Skills | 8 weeks
  Evaluation of static and dynamic balance performance using standardized balance tests pre- and post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Bingöl University Physical Education and Sports, Bingöl, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available to qualified researchers upon reasonable request, following publication of the main results. Data sharing will comply with ethical guidelines and privacy regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR